CLINICAL TRIAL: NCT03350555
Title: Validation of Clinical Use of Additioned Endoscopy in Endoscopic Retrograde Cholangiopancreatography
Brief Title: Clinical Trials to Validate the Use of Additioned Endoscopy in Endoscopic Retrograde Cholangiopancreatography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, Doctor of gastroenterology department, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Additioned Endocopy in ERCP
Record Dates: First submitted 2017-11-10; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: ERCP

STUDY DESIGN:
Intervention Model Description: One arm includes participants who will receive additioned endoscopy assisted ERCP, and the other arm includes participants who will not receive additioned endoscopy assisted ERCP.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP with additioned endoscopy (Experimental): This arm will include participants undergoing ERCP with assistance of additioned endoscopy.
  Interventions: Device: Additioned Endoscopy
- ERCP without additioned endoscopy (No Intervention): This arm will include participants undergoing ERCP without assistance of additioned endoscopy as negative controls.

INTERVENTIONS:
Device: Additioned Endoscopy — To evaluate the use of additioned endoscopy in ERCP treatment.
  Arms: ERCP with additioned endoscopy

SUMMARY:
Validation of clinical use of additioned endoscopy in Endoscopic Retrograde Cholangiopancreatography(ERCP) treatment.

DETAILED DESCRIPTION:
Investigators recently developed a device named additioned Endoscopy. The purpose of current clinical trial is to evaluate the use of additioned endoscopy in ERCP treatment, specifically in shortening the duration of ERCP operation and lowering incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* People who are indicated to ERCP treatment.

Exclusion Criteria:

* People who are not suitable for ERCP treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Duration of ERCP treatment | Duration of operation in each patient, ie. from beginning to the end of ERCP operation in each patient
  To test if additioned endoscopy will have impact on duration of ERCP treatment

SECONDARY OUTCOMES:
complications of ERCP treatment | up to 1 month after ERCP completion
  To test if additioned endoscopy will have impact on incidence of ERCP complications, including perforation, bleeding, post-ERCP pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No